CLINICAL TRIAL: NCT07119190
Title: Construction of a Perioperative Comprehensive Diagnosis and Treatment System for Lung Cancer in the Era of Neoadjuvant Immunotherapy
Brief Title: A Perioperative Comprehensive Diagnosis and Treatment System for Lung Cancer in the Era of Neoadjuvant Immunotherapy
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Collaborators: Beijing Municipal Health Commission (Other Government)
Responsible Party: Principal Investigator, Yang Fan, MD, Vice President, Peking University People's Hospital
Other Study IDs: BRWEP2024W034080200
Record Dates: First submitted 2025-07-15; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non-Small Cell Lung Cancer; Multiomics analysis; Tumor immune microenvironment; Radiomics; Pathological response; Immune-related adverse event; Nursing prehabilitation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — biopsy tissues and blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prospective cohort: Non-small cell Lung cancer patients receiving neoadjuvant immunotherapy and surgery

SUMMARY:
The goal of this study is to develop and refine an integrated minimally invasive care pathway for resectable lung cancer in the immunotherapy era, establishing a novel precision perioperative immunotherapy paradigm encompassing original techniques and clinical applications.

DETAILED DESCRIPTION:
Lung cancer remains the leading cause of cancer-related mortality in China and globally, imposing a substantial disease burden on society. Although comprehensive treatment strategies centered on surgery have improved patient outcomes, and perioperative immunotherapy-particularly immune checkpoint inhibitors-has profoundly reshaped the therapeutic landscape, significant knowledge gaps and critical challenges persist in this field. These challenges include uncertain beneficiary populations, poorly understood immune mechanisms, inaccurate efficacy prediction, difficult determination of resection margins, controversial efficacy assessment, and lack of effective early warning for adverse reactions.

This study will systematically identify biomarkers for early diagnosis and recurrence monitoring through multi-omic analysis of peripheral blood immune cell subsets and non-invasive liquid biopsies; investigate the tumor immune microenvironment's role in immunotherapy response mechanisms and predict treatment efficacy via multi-omic studies of tissue specimens; develop novel AI- and radiomics-assisted pathological assessment systems and prognostic prediction models; implement perioperative symptom assessment for timely identification of immune-related adverse events (irAEs) while conducting prehabilitation training for perioperative nursing care.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old;
2. NSCLC patients underwent radical surgical resection;
3. Adequate clinical-pathologic data, imaging data and follow-up data obtainable for multi-omics analysis;
4. Scheduled for or currently receiving neoadjuvant/perioperative immunotherapy.

Exclusion Criteria:

1. Histology of other malignant tumors, including concurrent malignant tumors of other organ systems;
2. Unresectable advanced disease (Stage IV) or locally advanced unresectable (Stage IIIC);
3. Pregnancy or lactation;
4. Insufficient sample quality;
5. Severe organ dysfunction (e.g. cardiac or renal insufficiency);
6. Other judgments by the Investigator that the patient should not participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who meet the eligibility criteria will be included consecutively
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2025-08-06 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response (pCR) | At surgery (typically 3-6 months post-treatment initiation)
  Pathologic Complete Response (pCR) is defined as the absence of residual tumor in both the primary lung tumor site and all sampled regional lymph nodes after neoadjuvant immunotherapy, confirmed through systematic pathological examination of the surgical specimen.

SECONDARY OUTCOMES:
Major Pathological Response (MPR) | At surgery (typically 3-6 months post-treatment initiation)
  Major Pathologic Response (MPR) is defined as the presence of ≤10% residual viable tumor cells in both the primary lung tumor site and sampled regional lymph nodes after neoadjuvant immunotherapy, confirmed through systematic pathological examination of the surgical specimen.
Objective Response Rate (ORR) | After two cycles or four cycles of neoadjuvant therapy (each cycle is 21 days).
  ORR is defined as the proportion of patients achieving either a complete response (CR; disappearance of all target lesions) or partial response (PR; ≥30% reduction in the sum of target lesion diameters) during or after neoadjuvant immunotherapy, as assessed by serial imaging (CT/PET-CT) using iRECIST criteria.
Recurrence-free Survival (RFS) | Through study completion, an average of 2 years
  Time from randomization to disease recurrence or death from any cause.
Overall Survival (OS) | Through study completion, an average of 2 years
  Time from randomization to death from any cause.
MRD (minimal residual disease) dynamics after neoadjuvant immunotherapy | Periprocedural and every three to six months post-treatment (up to three years)
  Postoperative dynamics of ctDNA-based MRD and timely detection of recurrence or metastasis in lung cancer patients receiving neoadjuvant immunotherapy.
Symptom Severity Score | Preoperative (T1: 2-4 weeks pre-surgery), postoperative (e.g., T3: 12-24 hours post-surgery, T5: 30 days post-surgery), and up to 90 days post-surgery.
  Assessment of perioperative symptom burden (e.g., pain, fatigue) using validated scales like the MDASI-C (M. D. Anderson Symptom Inventory) for lung cancer patients.
Immune-Related Adverse Event (irAE) Incidence | Periprocedural and up to 6 months post-treatment.
  Frequency and severity of adverse events (e.g., rash, colitis) related to immunotherapy, graded using standardized criteria like CTCAE (Common Terminology Criteria for Adverse Events).
Changes in PD-L1 expression (TPS) and TIL subpopulations (CD8+/FOXP3+ ratios, et al) before and after neoadjuvant immunotherapy | Periprocedural.
  PD-L1 expression (22C3 pharmDx assay; TPS ≥1% cutoff), multiplex immunofluorescence (CD8: clone C8/144B; FOXP3: clone 236A/E7) and multomoics analyses were performed on paired pre-/post-NAD biopsies.

CONTACTS AND LOCATIONS:
Overall Officials: Fan Yang, MD, Principal Investigator — Peking University People's Hospital

IPD SHARING:
Plan to Share IPD: Undecided